CLINICAL TRIAL: NCT02706301
Title: Pain Coping Skills Training for Colorectal Cancer Survivors With Pain and Distress
Brief Title: Pain Coping Skills for Colorectal Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00063330
Record Dates: First submitted 2016-03-08; First posted 2016-03-11 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer survivor; cancer pain; psychological distress; coping skills training; symptom management; cancer survivorship
MeSH Terms: conditions — Colorectal Neoplasms; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone-Based Coping Skills Training (CST) (Experimental): The CST condition will receive 5 sessions of a cognitive behavior theory-based protocol that teaches coping skills (e.g., relaxation, activity pacing/planning, cognitive restructuring) relevant to managing pain as well as psychological distress.
  Interventions: Behavioral: Telephone-Based Coping Skills Training (CST)
- Standard care control (No Intervention): The standard care control condition will receive resources and referrals related to survivorship health. This information will be provided to the participant during their initial survivorship care consult.

INTERVENTIONS:
Behavioral: Telephone-Based Coping Skills Training (CST)
  Arms: Telephone-Based Coping Skills Training (CST)

SUMMARY:
Colorectal cancer survivors experience long-term negative physical and psychosocial consequences of their disease. There is a critical need to develop novel behavioral interventions for improving colorectal cancer survivor outcomes. The investigators have developed a pain management intervention for colorectal cancer survivors that focuses on addressing both pain and psychological distress. Colorectal cancer survivors who endorse pain and comorbid psychological distress as a concern during a clinic-based survivorship care consult will be recruited. Participants will be randomized into either: Telephone-Based Coping Skills Training (CST) for pain and comorbid psychological distress or standard care. The CST condition will receive 5 sessions of a cognitive behavior theory-based protocol that teaches coping skills (e.g., relaxation, activity pacing/planning, cognitive restructuring) relevant to managing pain and psychological distress. The standard care control condition will receive resources and referrals related to managing survivorship health.

ELIGIBILITY:
Inclusion Criteria:

* >21 years old
* personal history of colorectal cancer
* finished active cancer treatment within the past 12 months
* reported pain as a concern as well as psychological distress on a National Comprehensive Cancer Network screener
* able to speak and read English
* able and willing to give informed consent

Exclusion Criteria:

* currently undergoing active cancer treatment
* have a major mental illness (e.g., schizophrenia)
* have a mental illness that is not being treated/controlled (e.g., bipolar disorder)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in Pain Severity assessed using the Brief Pain Inventory (BPI) | pre-treatment (baseline), post-treatment (approximately 8 weeks), 3-months post-treatment (approximately 20 weeks)
  Brief Pain Inventory (BPI)

SECONDARY OUTCOMES:
Change in Psychological Distress assessed using the Brief Symptom Inventory (BSI) | pre-treatment (baseline), post-treatment (approximately 8 weeks), 3-months post-treatment (approximately 20 weeks)
  Brief Symptom Inventory (BSI)
Change in Quality of Life assessed using the FACT-G, version 4.0 | pre-treatment (baseline), post-treatment (approximately 8 weeks), 3-months post-treatment (approximately 20 weeks)
  The Functional Assessment of Cancer Therapy - General (FACT-G), version 4.0
Change in Self-Efficacy for Pain Control assessed using the subscale of the Chronic Pain Self-Efficacy Scale | pre-treatment (baseline), post-treatment (approximately 8 weeks), 3-months post-treatment (approximately 20 weeks)
  Self-efficacy for pain management subscale of the Chronic Pain Self-Efficacy Scale

OTHER OUTCOMES:
Patient Satisfaction assessed using the Client Satisfaction Questionnaire 10-item version | Post-treatment (approximately 8 weeks)
  Client Satisfaction Questionnaire 10-item version.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A. Kelleher, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No